CLINICAL TRIAL: NCT01044537
Title: A Phase 1 Placebo-controlled Trial To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Single Escalating Oral Doses Of Pf-04937319 In Adult Subjects With Type 2 Diabetes Mellitus
Brief Title: A Trial To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Single Doses Of PF-04937319 In Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: B1621001
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: phase 1; safety and tolerability; PK; PD; type 2 diabetes mellitus; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — N,N-dimethyl-5-((2-methyl-6-((5-methylpyrazin-2-yl)carbamoyl)benzofuran-4-yl)oxy)pyrimidine-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): In each ascending-dose cohort, approximately 6 subjects will receive active treatment and 3 will receive placebo.
  Interventions: Drug: Placebo
- PF-04937319 (Experimental): In each ascending-dose cohort, approximately 6 subjects will receive active treatment and 3 will receive placebo. There will be approximately 6 dosing levels of PF-04937319
  Interventions: Drug: PF-04937319

INTERVENTIONS:
Drug: Placebo — Placebo to match PF-04937319 will be provided.
  Arms: Placebo
Drug: PF-04937319 — The initial planned dosing schedule is: 10, 30, 100, 200, and 400 mg, with one cohort to be determined. Doses shown may be adjusted upwards or downwards and may be adjusted to include intermediate doses. All doses will be administered as a single oral dose as a powder-in-capsule (PIC) formulation. PF-04937319 will be supplied as 10 mg and 80 mg (and potentially 1 mg) PIC.
  Arms: PF-04937319

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, pharmacokinetics, and pharmacodynamics of PF-04937319 following single escalating oral doses in adult subjects with Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
The purpose of this phase 1 study is to characterize the safety, tolerability, pharmacokinetics, and pharmacodynamics of PF04937319 following single escalating oral doses in adult subjects with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus who are taking stable doses of metformin only. Subjects treated with a sulfonylurea (SU) or a dipeptidyl peptidase-IV inhibitor (DPP-IVi) in combination with metformin may be eligible if washed off the SU or DPP-IVi to metformin only for a minimum of 4 weeks before dosing.
* Male and/or female subjects (females will be women of non childbearing potential) between the ages of 18 and 65 years, inclusive, with a body mass index (BMI) of 18.5 to 45.0 kg/m2 and C-peptide >0.8 ng/mL.
* Screening and Day -2 troponin I concentration </=0.05 ng/mL as measured by the Bayer Centaur Ultra assay.
* HbA1c >/=7% and </=11%. If the patient requires to be washed off an SU or DPP-IVi, the HbA1c limits will be >/=7% and </=9.5%.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Evidence or history of diabetic complications with significant end organ damage, eg, proliferative retinopathy and/or macular edema, creatinine clearance </=60 mL/min based on the Cockcroft-Gault equation, diabetic neuropathy complicated by neuropathic ulcers.
* History of stroke, transient ischemic attack, or myocardial infarction within the past 6 months. Additionally, history of coronary artery bypass graft or stent implantation, clinically significant peripheral vascular disease, or congestive heart failure (NYHA Classes II-IV). Furthermore, a current history of angina/unstable angina. Also, 12 lead electrocardiogram (ECG) demonstrating QTc >450 msec at screening, ECG findings suggestive of asymptomatic myocardial ischemia, or supine blood pressure >/=160 mm Hg (systolic) or </=100 mm Hg (diastolic).
* One or more self reported episodes of hypoglycemia within the last 3 months, or two or more self reported episodes of hypoglycemia within the last 6 months.
* Screening or Day -2 fasting (>/=8 hours) blood glucose, </=70 or >/=270 mg/dL, confirmed by a single repeat if deemed necessary.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Dedicated Phase 1, Phoenix, Arizona
  - West Coast Clinical Trials, LLC, Cypress, California
  - Elite Research Institute, Miami, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1621001&StudyName=A%20Trial%20To%20Assess%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%2C%20And%20Pharmacodynamics%20Of%20Single%20Doses%20Of%20PF-04937319%20In%20Subjects%20With%20T

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04937319 10 mg: Participants received single oral dose of PF-04937319 10 milligram (mg) capsule on Day 1.
- PF-04937319 30 mg: Participants received single oral dose of PF-04937319 30 mg (3 capsules of 10 mg) on Day 1.
- PF-04937319 100 mg: Participants received single oral dose of PF-04937319 100 mg (1 capsule of 80 mg and 2 capsules of 10 mg) on Day 1.
- PF-04937319 300 mg: Participants received single oral dose of PF-04937319 300 mg (3 capsules of 80 mg and 6 capsules of 10 mg) on Day 1.
- PF-04937319 480 mg: Participants received single oral dose of PF-04937319 480 mg (6 capsules of 80 mg) on Day 1.
- PF-04937319 640 mg: Participants received single oral dose of PF-04937319 640 mg (8 capsules of 80 mg) on Day 1.
- Placebo: Participants received single oral dose of placebo matched to PF-04937319 capsule on Day 1.
Period: Overall Study
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg | Placebo
Started | 6 | 6 | 6 | 6 | 5 | 5 | 16
Completed | 6 | 6 | 6 | 6 | 5 | 5 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 5 | 16 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (9.0) | 52.2 (8.8) | 52.0 (6.8) | 58.8 (4.6) | 55.0 (8.1) | 49.0 (10.0) | 53.7 (7.8) | 53.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 2 | 0 | 1 | 4 | 16
  Male | 2 | 4 | 3 | 4 | 5 | 4 | 12 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study medication and up to 10 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 up to 10 days after last dose of study medication (up to 11 days)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 5 | 16
participants
  AEs | 1 | 4 | 1 | 3 | 3 | 3 | 0
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Ratio of C-peptide Area Under Curve (C-peptide AUC) to Glucose Area Under Curve (Glucose AUC) After a Mixed Meal Tolerance Test (MMTT) on Day 1
Description: Ratio of area under the plasma C-peptide concentration-time curve from time 2 to 6 hrs (in terms of nanogram*deciliter*hour [ng*dL*hour]) to area under the plasma glucose concentration-time curve from time 2 to 6 hrs (in terms of milligram*milliliter*hour [mg*mL*hour]) was calculated. Linear trapezoidal method was used to compute AUC. The change in ratio from baseline (Day -1) was calculated at Day 1.
Time Frame: -46, -45.75, -45.5, -45, -44.5, -44, -43, -42 hours pre-dose on Day -1; 2, 2.25, 2.5, 3, 3.5, 4, 5, 6 hours post-dose on Day 1
Population: PD analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 of the PD parameters of interest. 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies participants evaluable at specified time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: (ng*dL*hour)/(mg*mL*hour)
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5 | 15
(ng*dL*hour)/(mg*mL*hour)
  Baseline (n= 5,6,6,6,5,5,15) | 0.02 (0.012) | 0.03 (0.014) | 0.03 (0.020) | 0.03 (0.009) | 0.03 (0.009) | 0.03 (0.009) | 0.03 (0.013)
  Change at Day 1 (n= 5,5,6,6,5,5,15) | 0.00 (0.002) | 0.00 (0.004) | 0.00 (0.013) | 0.01 (0.003) | 0.01 (0.005) | 0.01 (0.008) | 0.00 (0.005)

3. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration-time curve from zero to the last measured concentration (AUClast).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Population: Pharmacokinetic (PK) parameter analysis population included all enrolled participants who received study medication and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 5 | 5
nanogram*hour per milliliter | 475.2 (13) | 1362 (34) | 4418 (21) | 10640 (33) | 10830 (29) | 19970 (11)

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Population: PK parameter analysis population included all enrolled participants who received study medication and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 5 | 5
nanogram per milliliter (ng/mL) | 72.29 (25) | 124.9 (17) | 339.8 (34) | 756.6 (59) | 769.9 (50) | 1050 (24)

5. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 5 | 5
hour | 2.48 [1.95 to 3.00] | 2.50 [1.00 to 6.00] | 3.00 [1.95 to 8.00] | 3.50 [3.00 to 6.00] | 6.00 [1.92 to 6.00] | 7.98 [3.00 to 12.0]

6. Primary Outcome: Apparent Oral Clearance (CL/F)
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Population: PK parameter analysis population included all enrolled participants who received study medication and had at least 1 of the PK parameters of interest. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute (mL/min)
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 4 | 3
milliliter per minute (mL/min) | 344.8 (13) | 360.9 (37) | 364.4 (26) | 464.2 (40) | 690.3 (28) | 481.8 (10)

7. Primary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 4 | 3
liter | 154.0 (12) | 204.6 (42) | 254.4 (25) | 284.1 (76) | 379.2 (25) | 399.3 (23)

8. Primary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life (t1/2) is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 4 | 4
hour | 5.203 (0.74888) | 6.592 (0.79893) | 8.632 (3.3756) | 7.366 (2.4225) | 6.410 (1.0422) | 12.79 (6.3392)

9. Secondary Outcome: Percent Change From Baseline in Post-Prandial Glucose Area Under the Curve From Time 2 to 6 Hours (AUC [2-6]) After a Mixed Meal Tolerance Test (MMTT) on Day 1
Description: Percent change from baseline in post-prandial area under the plasma glucose concentration-time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC. Baseline value was the AUC (2-6) calculated on Day -1.
Time Frame: -46, -45.75, -45.5, -45, -44.5, -44, -43, -42 hrs pre-dose on Day -1; 2, 2.25, 2.5, 3, 3.5, 4, 5, 6 hrs post-dose on Day 1
Population: PD analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 of the PD parameters of interest. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 5 | 5 | 16
percent change | 8.58 (8.428) | -15.22 (8.887) | 4.96 (31.567) | -11.72 (8.350) | -10.81 (10.017) | -23.21 (10.207) | -0.45 (13.041)

10. Secondary Outcome: Percent Change From Baseline in Post-Prandial Insulin Area Under the Curve From Time 2 to 6 Hours (AUC [2-6]) After a Mixed Meal Tolerance Test (MMTT) on Day 1
Description: Percent change from baseline in post-prandial area under the plasma insulin concentration-time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC. Baseline value was the AUC (2-6) calculated on Day -1.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 5 | 5 | 14
percent change | 30.98 (21.327) | 10.72 (13.424) | 0.22 (26.086) | 2.03 (15.622) | 35.61 (28.235) | 9.30 (38.556) | 6.35 (25.752)

11. Secondary Outcome: Percent Change From Baseline in Post-Prandial C-peptide Area Under the Curve From Time 2 to 6 Hours (AUC [2-6]) After a Mixed Meal Tolerance Test (MMTT) on Day 1
Description: Percent change from baseline in post-prandial area under the plasma C-peptide concentration-time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC. Baseline value was the AUC (2-6) calculated on Day -1.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5 | 15
percent change | 14.10 (3.749) | -0.63 (14.664) | 1.79 (17.426) | 8.23 (8.101) | 21.13 (8.037) | 12.51 (19.188) | 6.09 (18.625)

12. Secondary Outcome: Change From Baseline in Ratio of Insulin Delta C30 to Glucose Delta C30 After a Mixed Meal Tolerance Test (MMTT) on Day 1
Description: Ratio of insulin delta C30 (in terms of milliunits*deciliter [mU*dL]) to glucose delta C30 (in terms of milligram*liter [mg*liter]) was calculated. The change in ratio from baseline (Day -1) was calculated at Day 1.
Time Frame: -46, -45.5 hrs pre-dose on Day -1; 2, 2.5 hrs post-dose on Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: (mU*dL)/(mg*Liter)
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 5 | 5 | 15
(mU*dL)/(mg*Liter)
  Baseline | 0.70 (0.627) | 4.59 (6.935) | 1.92 (2.759) | 0.77 (0.289) | 0.73 (0.265) | 0.85 (0.631) | 1.15 (0.798)
  Change at Day 1 | -0.04 (0.427) | -3.20 (7.093) | -0.81 (1.891) | 0.25 (0.090) | 1.89 (3.894) | 0.74 (0.675) | -0.05 (0.607)

13. Secondary Outcome: Change From Baseline in Ratio of C-peptide Delta C30 to Glucose Delta C30 After a Mixed Meal Tolerance Test (MMTT)
Description: Ratio of C-peptide Delta C30 (in terms of nanogram*deciliter [ng*dL]) to glucose delta C30 (in terms of milligram*milliliter [mg*mL]) was calculated. The change in ratio from baseline (Day -1) was calculated at Day 1.
Time Frame: -46, -45.5 hrs pre-dose on Day -1; 2, 2.5 hrs post-dose on Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: (ng*dL)/(mg*mL)
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5 | 15
(ng*dL)/(mg*mL)
  Baseline | 0.04 (0.034) | 0.16 (0.293) | 0.05 (0.064) | 0.03 (0.011) | 0.02 (0.008) | 0.05 (0.038) | 0.04 (0.023)
  Change at Day 1 | -0.01 (0.018) | -0.12 (0.283) | -0.02 (0.050) | 0.01 (0.006) | 0.13 (0.240) | 0.02 (0.029) | 0.00 (0.025)

14. Secondary Outcome: Change From Baseline in Ratio of Insulin Area Under Curve (Insulin AUC) to Glucose Area Under Curve (Glucose AUC) After a Mixed Meal Tolerance Test (MMTT) on Day 1
Description: Ratio of area under the plasma insulin concentration-time curve from time 2 to 6 hrs (in terms of milliunit*deciliter*hour [mU*dL*hour]) to area under the plasma glucose concentration-time curve from time 2 to 6 hrs (in terms of milligram*liter*hour [mg*liter*hour]) was calculated. Linear trapezoidal method was used to compute AUC. The change in ratio from baseline (Day -1) was calculated at Day 1.
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (mU*dL*hour)/(mg*liter*hour)
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 5 | 5 | 14
(mU*dL*hour)/(mg*liter*hour)
  Baseline (n= 5,5,6,6,5,5,14) | 0.24 (0.118) | 0.32 (0.257) | 0.48 (0.452) | 0.36 (0.142) | 0.29 (0.085) | 0.38 (0.310) | 0.34 (0.222)
  Change at Day 1 (n= 5,4,6,5,5,5,14) | 0.03 (0.036) | 0.10 (0.104) | -0.12 (0.235) | 0.04 (0.062) | 0.16 (0.104) | 0.10 (0.169) | 0.01 (0.071)

15. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf)
Description: AUCinf is the area under the plasma concentration versus time curve from time zero to extrapolated infinite time.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 4 | 3
nanogram*hour per milliliter | 483.3 (13) | 1385 (34) | 4570 (23) | 10770 (35) | 11590 (28) | 22130 (9)

ADVERSE EVENTS:
Arm/Group | PF-04937319 10 mg | PF-04937319 30 mg | PF-04937319 100 mg | PF-04937319 300 mg | PF-04937319 480 mg | PF-04937319 640 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/16
Other Adverse Events (participants affected / at risk) | 1/6 | 4/6 | 1/6 | 3/6 | 3/5 | 3/5 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04937319 10 mg (N=6) | PF-04937319 30 mg (N=6) | PF-04937319 100 mg (N=6) | PF-04937319 300 mg (N=6) | PF-04937319 480 mg (N=5) | PF-04937319 640 mg (N=5) | Placebo (N=16)
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Application site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.